CLINICAL TRIAL: NCT00384566
Title: The CAMERA Study: CArvedilol MEtoprolol Respiratory Assessment Investigator Trial
Brief Title: A Comparison of the Effect of Carvedilol and Metoprolol on Airways Tone in Patients With Heart Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: In order to join forces with another study already running which aims to answer the same question.
Sponsor: The Alfred (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Prof Henry Krum, Monash University / Alfred Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-03/04
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure; Chronic Obstructive Airway Disease
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Carvedilol; Metoprolol

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Carvedilol
- 2 (Active Comparator)
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Carvedilol — anit hypertensive medication
  Arms: 1
Drug: Metoprolol — Anti hypertensive medication
  Arms: 2

SUMMARY:
This study looks at the effect of two drugs (carvedilol and metoprolol) which are used for patients with CHF (chronic heart failure).

These agents are beta-blockers and, although effective in heart failure, may cause increases in airways tone and thus limit air getting into the lower parts of the lungs. Carvedilol is more active at blocking the receptor that opens up the airways and therefore theoretically may be more likely to reduce airways tone than metoprolol, although this has never been studied in patients with heart failure, and that is the purpose of the present study.

We are looking to enrol 45 patients with heart failure and mild obstruction to the flow of air in their lungs. Patients will be randomised to either carvedilol or metoprolol (standard doses). Following a minimum of 2 weeks of therapy of study medication the patient will undergo a study day involving an assessment of their lung function, an assessment of their heart failure, a "living with heart failure" questionnaire, blood tests and blood pressure and heart rate readings.

Patients will then be crossed over to the alternate medication. Following 2 weeks on the target dose the patient will undergo their second study day which will be the same as the first.

The results obtained from each study day will be compared.

ELIGIBILITY:
Inclusion Criteria:

* males and females over 18 years of age
* Documented CHF (NYHA class II-IV symptoms)
* Airflow obstruction defined as patients with symptomatic obstructive respiratory disease as manifest by any of the following Symptoms of wheeze, primarily attributed to airflow obstruction Requirement for intermittent or regular bronchodilator therapy FEV1 less than 70% predicted pre-salbutamol
* Confirmed written informed consent.
* Clinically indicated to receive β-blockade.
* No evidence of heart block on ECG.
* Patients will be in one of the following categories:

Currently on carvedilol Currently on Toprol-XL or Metoprolol tartrate Currently on bisoprolol Clinically indicated to receive β adrenoceptor blockade but not currently prescribed a β-blocker.

Exclusion Criteria:

* Women lactating, pregnant or of childbearing potential not using a reliable contraceptive method.
* Patients who had received an investigational new drug within the last 4 weeks.
* Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
* Laboratory parameters:

Creatinine >0.30 mmol/l Liver function tests 3x ULN

* Recent (<12 months) myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Respiratory function | Each study visit
NYHA class with the use of the 7 point scale (Packer). | Baseline, cross over, end of study
Minnesota "living with Heart Failure" questionnaire. | Baseline, cross over, end of study
U+E | Screening, cross over, end of study
BP and HR | every visit
plasma N-terminal pro-BNP | Screening, cross over, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, Professor, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia